CLINICAL TRIAL: NCT06494618
Title: The Effects of Botulinum Toxin Type a Injection Combined with RESWT in Lower Extremity Spasticity in Children with Cerebral Palsy
Brief Title: Effects of Botulinum Toxin Injection Combined with RESWT in Lower Extremity Spasticity in Children with Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, Bilinc Dugruoz Karatekin, M.D., Department of Physical Medicine and Rehabilitation, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP BTX ESWT
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy, Spastic
Keywords: cerebral palsy; spasticity; botulinum toxin injection; extracorporeal shockwave therapy
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Pediatric patients diagnosed with cerebral palsy who received botulinum toxin injection for lower extremity spasticity were randomized two groups. The first group will receive only conventional treatment after the injection, while the second group will receive extracorporeal shockwave therapy for injected muscles and their routine conventional therapy. The shock wave therapy is planned as 3 sessions per week, starting one week after the injection.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor were blinded to patients who received shockwave therapy and who did not received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum Toxin Injection and Conventional Therapy (No Intervention): The group received conventional therapy (such as stretching exercises) after Botulinum Toxin Type A Injection for spastic lower extremity muscle groups.
- Botulinum Toxin Injection and Shockwave Therapy (Active Comparator): The group received extracorporeal shockwave therapy conventional therapy (such as stretching exercises). Shockwave therapy is planned 3 sessions, starting first week after injection. It is planned to apply 1500 pulses, 4 hertz, 2 bars radial eswt to the injected spastic muscle groups in each session. The patients in this group will continue to their conventional therapy like the first group.
  Interventions: Device: Radial Extracorporeal Shockwave Therapy

INTERVENTIONS:
Device: Radial Extracorporeal Shockwave Therapy — 1500 pulses, 4 hertz, 2 bar radial extracorporeal shockwave therapy targeted muscle belly for botulinum toxin injected lower extremity muscle groups. 3 sessions were planned once a week, starting from first week after injection.
  Arms: Botulinum Toxin Injection and Shockwave Therapy

SUMMARY:
This study aimed to check and compare the effects of botulinum toxin injection combined with shock wave therapy versus botulinum toxin injection only for lower extremity spasticity in children with cerebral palsy

DETAILED DESCRIPTION:
20 pediatric patients diagnosed with cerebral palsy who received botulinum toxin type A injection for lower extremity spasticity were divided into two groups. The first group will receive only conventional treatment after the injection, while the second group will receive extracorporeal shockwave therapy for injected muscles. The shock wave therapy is planned as 3 sessions per week, starting one week after the injection. Patients will be compared in terms of MAS scores, MTS scores, passive joint range of motion, modified timed up and go test, pain scores, (faces pain scale-revised) and Goal Attainment Scaling scores. Patients will be evaluated 1 week, 1 month and 3 months after the injection with pre-injection data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cerebral palsy.
* Spasticity in at least one of the lower extremity muscle groups.
* No contraindications to shockwave therapy.
* Applied Botulinum Toxin Type A injection for at least one spastic muscle of lower extremity.
* Agreed to participate to study (patient/primary caregiver)

Exclusion Criteria:

* Surgery history within the last year of the muscle to be injected and treated
* Having uncontrolled epilepsy.
* Having infection
* Coagulopathy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Modified Aschworth Scale | 3 months (before injection, first week, first month and third month after injection.)
  Scoring system used to evaluate spasticity. Spasticity scored as 0, 1, 1+, 2, 3, 4.
Modified Tradiue Scale | 3 months (before injection, first week, first month and third month after injection.)
  Scoring system used to evaluate spasticity. Spasticity scored as 0,1,2,3,4.
Modified Timed Up and Go Test | 3 months (before injection, first week, first month and third month after injection.
  The test for evaluate the functionality of pediatric patients with cerebral palsy. Only one chair and a surface for the patient to walk three meters are required. The time it takes for the patient to get up from the chair, walk the specified distance and sit back in the chair is recorded.
Facies Pain Scale Revised | 3 months (before injection, first week, first month and third month after injection.)
  The scale for evaluate the pain level of pediatric patients. Chosen faces are scored 0, 2, 4, 6, 8, or 10, counting left to right, so "0" equals "No pain" and "10" equals "Very much pain."
Passive Range of Motion | 3 months (before injection, first week, first month and third month after injection.)
  Goniometric measurement of the range of motion of the joint of the injected muscle
Goal Attaintment Scale | 3 months (before injection, first week, first month and third month after injection.)
  The method of scoring the extent to which patient's individual goals are achieved in the course of intervention. GAS comprises of goals divided into a 5-point scale from -2 to +2.
  Achievement of goal = 0 Achieved somewhat more than expected outcome = +1 Achievement of much more than expected goal = +2 Achievement of somewhat less than expected goal = -1 Achievement of much less than expected goal = -2

CONTACTS AND LOCATIONS:
Overall Officials: Belgin Erhan, Assoc. Prof., Study Director — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No